CLINICAL TRIAL: NCT04656184
Title: A Randomized Phase III Multicenter Trial Comparing the Efficacy and Safety of Anakinra Versus Intravenous Immunoglobulin (IVIG) Retreatment, in Patients With Kawasaki Disease Who Failed to Respond to Initial Standard IVIG Treatment
Brief Title: A Trial Comparing the Efficacy and Safety of Anakinra Versus Intravenous Immunoglobulin (IVIG) Retreatment, in Patients With Kawasaki Disease Who Failed to Respond to Initial Standard IVIG Treatment
Acronym: ANACOMP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P200009
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Kawasaki Disease
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome | interventions — Interleukin 1 Receptor Antagonist Protein; Immunoglobulins, Intravenous

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KINERET (Experimental): The patients will receive anakinra, an analogue of the IL-1 receptor antagonist, at a starting dose of 4 mg/kg. If patients are still febrile with 12 hours (H12) of treatment, they will receive a supplementary dose of 2 mg/Kg; otherwise, they will remain at a starting dose of 4 mg/kg. If they are still febrile at H24, they will receive a dose of 8mg/kg; otherwise, they will maintain their dose of 6 mg/kg. Patients with temperature <38°C at any point between initiation and day 14, but who develop secondary fever due to KD could have further escalation dose of anakinra until a maximum dose of 8mg/Kg. Patients will receive anakinra during 14 days independently of the period of escalation dose if any. After the last escalation dose, if any necessary, the primary criteria will be measured. Patients not responding to anakinra will follow usual standard care and will complete information related to all the study visits
  Interventions: Drug: ANAKINRA
- Intravenous Immunoglobulin (Active Comparator): The patients will receive a standard therapy, IVIG infusion of 2g/kg, and their treatment will follow usual standard care. Patients in the IVIG treatment will complete information related to the study visits.
  Interventions: Drug: Intravenous immunoglobulin

INTERVENTIONS:
Drug: ANAKINRA — The patients will receive anakinra, an analogue of the IL-1 receptor antagonist, at a starting dose of 4 mg/kg. If patients are still febrile with 12 hours (H12) of treatment, they will receive a supplementary dose of 2 mg/Kg; otherwise, they will remain at a starting dose of 4 mg/kg. If they are still febrile at H24, they will receive a dose of 8mg/kg; otherwise, they will maintain their dose of 6 mg/kg. Patients with temperature <38°C at any point between initiation and day 14, but who develop secondary fever due to KD could have further escalation dose of anakinra until a maximum dose of 8mg/Kg. Patients will receive anakinra during 14 days independently of the period of escalation dose if any. After the last escalation dose, if any necessary, the primary criteria will be measured. Patients not responding to anakinra will follow usual standard care and will complete information related to all the study visits
  Other Names: Kineret
  Arms: KINERET
Drug: Intravenous immunoglobulin — The patients will receive a standard therapy, IVIG infusion of 2g/kg, and their treatment will follow usual standard care. Patients in the IVIG treatment will complete information related to the study visits.
  Arms: Intravenous Immunoglobulin

SUMMARY:
Kawasaki disease (KD) is the most frequent vasculitis in younger children <5years, and the first cause of acquired ischemic myocardiopathy in childhood. Exceptionally, KD may cause early death during the acute phase by myocardial infarction, but may compromise the long-term cardiovascular outcome by accelerating atherosclerotic disease.

The incidence of KD is high in far-Eastern countries and Hawaii but KD is relatively rare in other regions (10/100000 children <5years in northern Europe) which makes it difficult to develop research on these rare population.

Early recognition and treatment by intravenous immunoglobulins (IVIG) influences the prognosis positively. IVIG are the standard of care and decrease significantly the risk of coronary aneurysms. However, despite a first infusion of IVIG, 20% of KD patients remain febrile and have high risk of coronary vasculitis. Recent Japanese research group assessed additional cyclosporine treatment in first line KD treatment but failed preventing relapse. To date there is no agreement for a more effective second line treatment.

Based on the auto-inflammatory pattern of KD, the investigators hypothesize that anti IL-1 blocking agents could bring a rapid and sustained effect on systemic and coronary inflammation in patients with KD.

Our hypotheses are:

1. Anakinra treatment may reduce the early and long-term mortality of patients with Kawasaki Disease (KD), by a rapid and sustained effect on vascular inflammation.
2. The safety of anakinra is good, as the drug has a very short half-life, which allows its rapid withdrawal in case of serious adverse event.

The use of anakinra is not associated with the risk of contamination by infectious agents, which remain even minimal, a possibility with the use of IVIG.

DETAILED DESCRIPTION:
It is a multicentric national randomized controlled, parallel-group in a 1:1 ratio, open labelled trial of superiority.

The main objective is to compare the efficacy of Anakinra (Interleukin 1 receptor type 1 - receptor antagonist) with 2nd IVIG infusion, in second line, on fever in patients with KD, who failed to respond to one infusion of IVIG(standard treatment).

The main criterion-evaluating efficacy in both groups is: the patient must reach a body (axillary (+0.5°C), tympanic, oral) temperature <38˚C within 2 days after initiation of treatment (i.e. a binary outcome: success/failure).

The secondary objectives are to compare Anakinra with IVIG retreatment in terms of:

* Efficacy on fever at 72h
* Efficacy on disease activity
* Efficacy on KD symptoms
* Efficacy on coronary lesions (e.g.: dilatation and aneurysm)
* Efficacy on inflammation
* Safety and tolerability Secondary End Points (linked with the secondary objectives)

To compare Anakinra with IVIG retreatment in terms of:

* Temperature <38˚C within 3 days (72h) after initiation of treatment
* Decrease of the CRP values from baseline to day 30(CRP<6 mg/L at day 30)
* Reduction in physician assessment of disease activity, on a 10 points scale, of at least to 50% between baseline and day 14.
* Reduction in patient's parent's assessment of disease activity, on a 10 points scale, of to at least 50% between baseline and day 14.
* Resolution of coronary abnormalities; i.e worst Z score <2.5, by echocardiogram if present at day 45.
* Adverse events: pain/redness at injection site, bacterial infection hepatitis, macrophage activation syndrome, severe neutropenia,
* Monitoring of adverse events

  * Physical examination: Complete clinical exam will be performed at each visit to detect symptoms of KD (rash, cervical nodes, mucous lesions, extremities, GI, pulmonary, cardio vascular, neurologic and muscular/joint evaluation) and possible associated morbidity: e.g. concomitant infection
  * Local tolerability of injections: will be evaluated by physician from V2 to V8: pain, redness, swelling, induration, itching, haemorrhage, (and quoted from none, mild, moderate, severe)
  * Vital signs and body measurements: at each visit: V1 to V9. The body temperature will be measured daily until d30. Parents will receive a follow-up booklet..
  * Laboratory evaluations: hematologic, hepatic and renal assessment will be followed

Group 1: KINERET:

KINERET® in the form of prefilled syringe with 100 mg of anakinra per 0.67 ml (150 mg/mL) and adapted to paediatric population, in pack sizes of 7. Patients in group I, will receive a starting dose of anakinra is 4 mg/kg at visit D1 (or day 0, if possible). During visits D1 and D2, if patients are still febrile with 12 hours (H12) of treatment, they will receive a supplementary dose of 2 mg/Kg; otherwise, they will remain at a starting dose of 4mg/kg. If they are still febrile at H24, they will receive a dose of 8mg/kg; otherwise, they will maintain their dose of 6 mg/kg. Patients with temperature <38°C at any point between initiation and day 14, but who develop secondary fever due to KD could have further escalation dose of anakinra until a maximum dose of 8mg/Kg.

Group 2: IVIG Immunoglobulins concentrates used for the ANACOMP study should be preferably the specialty PRIVIGEN® 100mg/mL (=10g of human immunoglobulins) solute for intravenous infusion, manufactured by CSL Behring (Commonwealth Serum Laboratories). Other presentations in mL (25, 50, 200, 400 exist corresponding to respectively 2.5g, 5g, 20, and 40g of immunoglobulins). Patients in group II, will receive one infusion of 2g/kg of intravenous Immunoglobulins at visit D1 (or day 0, if possible)

ELIGIBILITY:
Inclusion Criteria:

* Children, male and female, from 3 months to <18 years old
* Patient ≥ 5 kg
* Patient with KD according to the American Heart Association definition for complete or incomplete KD. (Fever ≥ 5 days (or at least 3 days if KD with American Heart Association criteria since the third days of fever) and ≥ 4 of 5 main clinical signs: modification of the extremities, polymorphic exanthema, and bilateral bulbar not exudative conjunctivitis, erythema of the lips or oral cavity, and cervical lymph nodes usually unilateral > 1.5 cm in diameter.
* Patients who failed to respond to the standard therapy of KD, e.g. Persistence or recrudescence of fever ≥ 38°C, 48 hours after the infusion of 2g/kg of IV Ig. Patients may be screened 24h after the end of the first infusion if they remain febrile 24h after the end of the first infusion.
* Patient, parents or legal guardian's written informed consent is required
* Patient with health insurance (SS or CMU).
* Efficient contraception for the duration of participation in the research for childbearing aged women

Exclusion Criteria:

* Preterm and neonates, pregnancy, pregnancy and breast feeding
* Suspicion of another diagnosis
* Patient with overt concomitant bacterial, viral or fungal infection
* Patient previously treated with steroids and/or another biotherapy
* Patient with increased risk of tuberculosis infection
* Recent tuberculosis infection or with active tuberculosis
* Patient with any type of immunodeficiency or cancer
* Patients with severe renal impairment (CLcr < 30 ml/minute)
* Patients with hepatic insufficiency
* Patients with neutropenia (ANC<1.5 x109/l)
* Patients included in another interventional protocol
* Patient under the following treatments:
* Preventive Antipyretics (paracetamol, NSAIDs other than aspirin 30-50mg/kg given for purpose of KD inflammation), as long as the patient receives the study medication
* Immunosuppressive medications given in a period less than twice of their half-life prior the patient receives the study medication (systemic steroids, cyclosporine, tacrolimus, azathioprine, cyclophosphamide, interferon, mycophenolate, other anti-IL-1, anti IL-6, anti CD20 and anti TNF (Tumor Necrosis Factor)), plasmapheresis)
* Hypersensitivity to anakinra or excipients (citric acid, sodium chloride, disodium EDTA (Ethylene Diamine Tetra Acetic), polysorbate 80, sodium hydroxide, in water for injection)
* Hypersensitivity to IV Ig, or excipients (L-proline and water for injection), hypersensitivity to human normal immunoglobulin, in particular if the patient have anti-IgA antibodies (IgA: Immunoglobulin A)
* Patients with type I or II hyperprolinemia
* Live vaccines within 1 month prior to enrollment
* Hypersensitivity to anakinra or to immunoglobulins or to excipients of Kineret® or Privigen® or to E.coli proteins
* Contraindication for administration of anakinra or IVIG listed in the Summary of Products Characteristics (SmPC) of Kineret® and Privigen®
* Ongoing or recent use of any other medication Known inhibitors/inducers of cytochrome P450 as listed on the link below: http://medicine.iupui.edu/clinpharm/ddis/main-table

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Fever | 48 hours
  The main criterion-evaluating efficacy in both groups is: the patient must reach a body (axillary (+0.5°C), tympanic, oral) temperature <38˚C within 2 days after initiation of treatment (i.e. a binary outcome: success/failure).

SECONDARY OUTCOMES:
Fever | day 3, day 4, day 6, day 7, day 14, day 30, day 45, day 60
  a body (axillary (+0.5°C), tympanic, oral) temperature >38˚C
CRP | day 3 (or day 4) day 7, day 14, day 30 and day 45.
  Decrease of the CRP values
Disease activity (physician assessment) | day 2, day 3, day 4, day 6, day 7, day 14, day 30, day 45, day 60
  Reduction in physician assessment of disease activity, on a 10 points scale, of at least to 50%
Disease activity (patient's parent's assessment) | day 2, day 3, day 4, day 6, day 7, day 14, day 30, day 45, day 60
  Reduction in patient's parent's assessment of disease activity, on a 10 points scale, of to at least 50%
Coronary abnormalities | Day 45
  Resolution of coronary abnormalities; i.e worst Z score <2.5, by echocardiogram if present
Safety and tolerability | From baseline to day 60 (day 2, day 3, day 4, day 6, day 7, day 14, day 30, day 45 and day 60)
  Adverse events: pain/redness at injection site, bacterial infection hepatitis, macrophage activation syndrome, severe neutropenia,

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bicêtre, Le Kremlin-Bicêtre, Val De Marne, France

IPD SHARING:
Plan to Share IPD: Undecided